CLINICAL TRIAL: NCT02878434
Title: Fertility Preservation in Young Women With Cancer: an International Registration Study From the International Network on Cancer, Infertility and Pregnancy (INCIP)
Brief Title: Fertility Preservation in Young Women With Cancer
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: NKI-AvL (Unknown); Medical University of Vienna (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); N.N. Blokchin NMRCO (Unknown)
Responsible Party: Principal Investigator, Frederic Amant, MD PhD, University Hospital, Gasthuisberg
Other Study IDs: INCIP Fer
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Fertility
Keywords: Cancer; Fertility; Pregnancy; Chemotherapy; Radiotherapy; Long term; Follow up
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group
- control group

SUMMARY:
The researchers aim to record the incidence, treatment and long term follow up of fertility preserving cancer treatment. Both the oncological and fertility outcome are recorded.

Study population: All patients with a cancer for whom a fertility preserving cancer treatment is applied. The results of the study population are compared to young women undergoing standard cancer treatment.

DETAILED DESCRIPTION:
Cancer is the second leading cause of death during the reproductive years. The long term survival improves for most cancers, reaching 80% for pediatric cancer and more than 70% for cancers in adults between 20 and 49 years of age. Early detection and improvements in cancer treatment contribute to these figures. As a result, quality of life of which preservation of fertility is one aspect, becomes more important. Fertility may however be influenced by surgery and by the gonadotoxic effects of chemo and/or radiotherapy. Therefore, fertility sparing treatments are offered to young patients in order to maintain the wish to conceive after cancer treatment. This however is associated with deviation of standard treatment and many different strategies are applied among different centers. In addition, there is a lack of studies investigating the oncological safety of these fertility sparing treatment protocols. The results of this study will enable us to better inform clinicians and patients on the efficacy of fertility sparing cancer treatment.

Objective:

To record the incidence, treatment and long term follow up of fertility preserving cancer treatment. Both the oncological and fertility outcome are recorded.

Study design: International multicentre prospective observational trial

Study population: All patients with a cancer for whom a fertility preserving cancer treatment is applied. The results of the study population are compared to young women undergoing standard cancer treatment.

Main study parameters/endpoints:

Registration of cancer diagnosis, treatment and outcome. Both the oncologic and fertility outcome is registered.

All patients receive fertility sparing cancer treatment on their specific request.

ELIGIBILITY:
Inclusion Criteria:

* Young women who want to preserve their fertility during cancer treatment. Patients need to give their signed and written informed consent to participate in the study.

Exclusion Criteria:

* Mentally disabled or significantly altered mental status that would prohibit the understanding and giving of informed consent

Ages: 0 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All women diagnosed with cancer for whom a fertility preserving cancer treatment is applied will be considered for inclusion.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Fertility Outcome | 10 years
  pregnancy rate

SECONDARY OUTCOMES:
Oncological Outcome | 5 years
  Recurrence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Amant, MD, PhD, Principal Investigator — UZ Gasthuisberg & KU Leuven, Belgium
Locations (2):
- UZ Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium
- The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This site provides background information on the problem of cancer in pregnancy and cancer and fertility — http://www.cancerinpregnancy.org

DOCUMENTS (4):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02878434/Prot_000.pdf
  • Informed Consent Form: adult (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02878434/ICF_001.pdf
  • Informed Consent Form: child -18y (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02878434/ICF_002.pdf
  • Informed Consent Form: parent for child -18y (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02878434/ICF_003.pdf